CLINICAL TRIAL: NCT03710798
Title: Effect of an Low Carbon High Fat Diet on Pain- and Quality of Life in Patients With Lipedema
Acronym: LIPODIET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helse Nord-Trøndelag HF (Other)
Collaborators: St. Olavs Hospital (Other); University of Oslo (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018/307
Record Dates: First submitted 2018-10-16; First posted 2018-10-18 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Lipedema; Obesity, Morbid
Keywords: Diet, ketogenic; Pain; Quality of Life; Body Composition; Body Fat Distribution
MeSH Terms: conditions — Lipedema; Obesity, Morbid; Pain | interventions — Diet, Ketogenic

STUDY DESIGN:
Intervention Model Description: prospective observational study with a diet intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Low carbohydrate high fat diet (Experimental): Low carbohydrate high fat (LCHF) diet
  Interventions: Dietary Supplement: Low carbohydrate high fat diet

INTERVENTIONS:
Dietary Supplement: Low carbohydrate high fat diet — Energy balanced low carbohydrate high fat diet during 6 weeks. Then 6-week reintroduction of a healthy normal diet
  Other Names: ketogenic diet

SUMMARY:
Lipedema is a chronic disease with unproportional, symmetrical fat accumulation in the lower extremities. Patients experience pain in affected areas, and reduced quality of life. Today's treatment is physiotherapy and surgery (liposuction). Recent research shows that ketogenic-diet with low carbohydrate, high fat (LCHF) conant can lead to reduced pain, increased quality of life and change in body composition. Goals: Investigate the effect of LCHF diet on pain, quality of life and body composition.

ELIGIBILITY:
Inclusion Criteria:

* weight stable over the last three months (+ 2-3 kg)
* not currently dieting to loose weight.
* willing to meet for weekly follow-ups during the intervention and the reintroduction of a regular diet.
* sign an informed consent before entering the study.

Exclusion Criteria:

* pregnant or breast feeding
* history of infectious diseases
* medication known to affect obesity
* enrolment in any other obesity treatment
* have had a bariatric surgery
* history of psychological disorders
* mentally disabled
* not mastering a Scandinavian language
* having a malign disease or any disease that leads to dietary advice that is not consistent with intervention advices in the study

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-01-10 (Actual); Study Completion 2019-01-10 (Actual)

PRIMARY OUTCOMES:
Lymphedema Quality of Life questionnaire | 6 weeks
Pain indicated on a visual analog scale | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bodil Landstad, prof, Study Director — Norwegian University for Science and Technology
Locations (1):
- Obesity Clinic, St Olavs Hospital, Trondheim, Norway

IPD SHARING:
Plan to Share IPD: Undecided